CLINICAL TRIAL: NCT01138566
Title: Clinical Significance and Optimal Treatment of Community-onset Urinary Tract Infections Caused by Extended-spectrum β-lactamase and/or AmpC β-lactamase Producing Enterobacteriaceae
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Other Study IDs: IISP37925
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Tract Infections
Keywords: community-onset urinary tract infections caused by Enterobacteriaceae
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ESBL- and/or AmpC-(+) or (-)

SUMMARY:
The purposes of this study are:

1. To estimate the prevalence of extended spectrum β-lactamase (ESBL) and/or AmpC among Enterobacteriaceae which cause community-onset urinary tract infections (UTIs)
2. To collect the background, risk factors and clinical outcome of patients with community-acquired uropathogenic condition related to Enterobacteriaceae (both ESBL, AmpC- and non ESBL and/or AmpC producing) after receive different antibiotic regimens.
3. To develop a scoring system to early identify patients at risk of being infected with ESBL- and/or AmpC-producing Enterobacteriaceae by comparing the risk factors for community-onset UTIs caused by ESBL- and/or AmpC-positive against non ESBL -and/or AmpC Enterobacteriaceae
4. To demonstrate the efficacy and safety of ertapenem for the empiric treatment of community-onset UTIs in patients at risk for ESBL- and/or AmpC-producing organism.

The study hypothesis (i) Patients infected with community-acquired uropathogenic ESBL- and/or AmpC-producing Enterobacteriaceae who receive regimens other than carbapenems have a worse outcome.

(ii) There are certain risk factors predicting the acquisition of community-onset UTIs caused by ESBL- and/or AmpC-producing Enterobacteriaceae.

(iii) The use of ertapenem is an effective and safe empirical therapy compared with other agents for community-onset UTIs caused by ESBL- and/or AmpC-producing Enterobacteriaceae.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who admitted to the Taipei Veterans General Hospital with the diagnosis of community-onset UTI caused by Enterobacteriaceae will be eligible for inclusion in this study if hospitalization for parental antimicrobial therapy is required

Exclusion Criteria:

* pregnancy or lactation in women,
* history of serious allergy or intolerance to study drug therapy (patients with a history of mild rash to β-lactams could be enrolled),
* complete obstruction of the urinary tract,
* peri-nephritic or intrarenal abscess, prostatitis, any rapidly progressive disease or terminal illness,
* immuno-compromising illness or immuno suppression therapy, the need for concomitant antimicrobials in addition to study therapy,
* a baseline pathogen resistant to study drug,
* treatment with a systemic antimicrobial agent for >24 h within 72 h prior to enrolment, or absolute neutrophil count <1000/mm3.
* Men with a history or physical findings suggestive of acute or chronic prostatitis will also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who admitted to the Taipei Veterans General Hospital, a 2900-bed tertiary-care teaching hospital located in Taipei, Taiwan, with the diagnosis of community-onset UTI caused by Enterobacteriaceae
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Vterans General Hospital, Taipei, Taiwan